CLINICAL TRIAL: NCT00380315
Title: Therapeutic Confirmatory Clinical Trial to Evaluate the Safety and Efficacy of AG1321001 Capsule as an Anti-Tussive Agent in Cough Patients: Double Blinded, Randomized, Placebo and Active Rug Comparative, Parallel Designed Phase III Study
Brief Title: Therapeutic Confirmatory Clinical Trial to Evaluate the Safety and Efficacy of AG1321001 in Chronic Cougher
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ahn-Gook Pharmaceuticals Co.,Ltd (Industry)
Responsible Party: Jung Hoon Han / Project Development Team
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AG1321001_P302
Record Dates: First submitted 2006-09-21; First posted 2006-09-25 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-06

CONDITIONS: Cough
Keywords: Cough; Chronic bronchitis; PNDs; Post Nasal Drip syndrome; GERD; gastroesophageal reflux disease; bronchiectasis
MeSH Terms: conditions — Cough; Bronchitis, Chronic; upper airway cough syndrome; Gastroesophageal Reflux; Bronchiectasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

INTERVENTIONS:
Drug: AG1321001(drug)

SUMMARY:
This study is for therapeutic confirmation of AG1321001 to evaluate the safety and efficacy as an anti-tussive agent in cough patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult between the ages of 18 and 70.
2. Patient who has cough symptom caused by following diseases: chronic bronchitis, bronchiectasis, gastroesophageal reflux disease, postnasal drip syndrome caused by rhinitis, sinusitis, rhinopharyngitis, rhinolaryngitis.
3. Patient requiring internal treatment due to cough symptom, who has coughing more than 3 weeks.
4. patient who will continue to cough more than 1 week.(by physician's judgment)
5. Patient who decided to participate in this clinical trial at his(her) own will and agreed in written letter of consent.
6. Patient who is trustworthy, ready for cooperation and observing the restrictions during the trial period.

Exclusion Criteria:

1. Patient who is accompanied by the seriously abnormal symptom in respiratory system, such as Acute infectious Pulmonary Disease, Tuberculosis.
2. Patient who has clinical history of sensitivity to Xanthine drug.
3. Patient who has Peptic Ulcer or Asthma (Except Cicatrix)
4. Patient whose liver or kidney function is seriously abnormal: Including the cases of sGOT, sGPT, bilirubin and blood creatinine value exceeding twice of their upper normal limit.
5. Patient whose heart function is abnormal: including the case of showing abnormal EKG test value that is clinically significant.
6. Patient who has experience to have participated in other clinical trial within two months before starting the trial.
7. Pregnant woman, lactating woman.
8. patient who has convulsion or alcoholism.
9. patient who take medicines which can not use combination with AG1321001.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2006-03; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Cough severity, Cough specific Quality of Life

SECONDARY OUTCOMES:
Daily cough symptom, Cough frequency

CONTACTS AND LOCATIONS:
Overall Officials: Young-hwan Kim, MD, PhD, Study Chair — Seoul National University Hospital, Seoul, 110-744, Korea, Republic of; Choon-Taek Lee, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital, Sungnam, Korea, Republic of; Hee-Soon Chung, MD, PhD, Principal Investigator — Seoul National University Boramae Hospital, Seoul, 156-707, Korea, Republic of; Ki-suk Jung, MD, PhD, Principal Investigator — Hallym University Sacred Heart Hospital, Anyang, Kyunggi, 430-070, Korea, Republic of; Joon Chang, MD, PhD, Principal Investigator — Severance Hospital, Seoul, 120-752, Korea, Republic of; Chul-min Ahn, MD, PhD, Principal Investigator — Yongdong Sevenrance Hospital, Seoul, 135-720, Korea, Republic of
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- See also: Related Info — http://www.ahn-gook.com